CLINICAL TRIAL: NCT00002401
Title: An Open-Label Randomized Study of Delavirdine Mesylate (DLV, Rescriptor) in Triple and Quadruple Combinations With Zidovudine (ZDV), Indinavir (IDV), and Lamivudine (3TC) in HIV-1 Infected Individuals
Brief Title: A Study of Delavirdine Used Together With Other Anti-HIV Drugs in HIV-Infected Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pharmacia and Upjohn (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 228F; 0074
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-01

CONDITIONS: HIV Infections
Keywords: HIV-1; Zidovudine; HIV Protease Inhibitors; Lamivudine; Indinavir; RNA, Viral; Delavirdine; Reverse Transcriptase Inhibitors; Viral Load
MeSH Terms: conditions — HIV Infections | interventions — Indinavir; Delavirdine; Lamivudine; Zidovudine

INTERVENTIONS:
Drug: Indinavir sulfate
Drug: Delavirdine mesylate
Drug: Lamivudine
Drug: Zidovudine

SUMMARY:
The purpose of this study is to see if it is safe and effective to give delavirdine (DLV) in combination with two or three other drugs to HIV-infected patients. The drugs to be used in combination with DLV are zidovudine (ZDV), indinavir (IDV), and lamivudine (3TC).

DETAILED DESCRIPTION:
In this open-label pilot study, patients are randomized to 1of the following 4 arms for 24 weeks:

Arm 1 (40 patients): DLV plus ZDV plus IDV. Arm 2 (40 patients): DLV plus IDV plus 3TC*. Arm 3 (40 patients): DLV plus ZDV plus IDV plus 3TC. Arm 4 (40 patients): ZDV plus IDV plus 3TC.

* Dose determined by body weight. Patients may opt to continue on study for 24 additional weeks at the discretion of the investigator.

ELIGIBILITY:
Inclusion Criteria

Prior Medication:

Allowed:

Less than 1 month prior treatment with zidovudine.

Exclusion Criteria

Prior Medication:

Excluded:

* Prior indinavir.
* Prior lamivudine.
* Prior protease inhibitors.
* Prior non-nucleoside reverse transcriptase inhibitors.
* 1 month or more prior zidovudine.

  1. HIV-1 positive.
* CD4 coun tis above 50.
* HIV-1 RNA levels greater than 20,000.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 160

CONTACTS AND LOCATIONS:
Locations (1):
- Pharmacia & Upjohn, Peapack, New Jersey, United States